CLINICAL TRIAL: NCT03695822
Title: Far Eastern Memorial Hospital
Brief Title: Impact of Beta-3 Agonist on Psychological Distress and Blood Flow of the Bladder in Women With Overactive Bladder Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: I did not pass the 2018 Ministry of Science and Technology research project subsidy, so I applied for the project to close the case.
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107009-F
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-05

CONDITIONS: Overactive Bladder Syndrome
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mirabegron (Experimental): OAB female patients who will receive beta-3 agonist (mirabegron 2 mg) treatment
  Interventions: Drug: Mirabegron 25mg

INTERVENTIONS:
Drug: Mirabegron 25mg — The aim of this study is to elucidate the impact of mirabegron on psychological distress, bladder blood flow and c reactive protein.

SUMMARY:
We will get the impact of mirabegron on psychological distress, urethra and bladder blood flow and c reactive protein.

DETAILED DESCRIPTION:
Background/Purpose: Pharmacologic treatments for female overactive bladder syndrome (OAB) include antimuscarinics and beta-agonist. Similar efficacy has been reported between antimuscarinics and beta-agonist. Antimuscarinics has been found to be beneficial for patients with psychological distress. However, the impact of mirabegron on psychological distress in female OAB remains unknown. In addition, some animal studies found that beta-3 agonist can improve arterial blood flow, bladder ischemia and might improve bladder function; however, there is still lack of human study. Besides, c reactive protein was found to be elevated in female OAB. Nonetheless there is no study mentioning about the impact of mirabegron on c reactive protein. Thus, the aim of this study is to elucidate the impact of mirabegron on psychological distress, bladder blood flow and c reactive protein.

ELIGIBILITY:
Inclusion Criteria:

* All OAB female patients
* >20 years

Exclusion Criteria:

* Allergy to mirabegron, urinary tract infections

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Brief symptom rating scale | 12 weeks
  The Brief symptom rating scale (BSRS) includes the following dimensions of psychopathology: somatic symptoms, obsessive-compulsive symptoms, interpersonal sensitivity, depressive symptoms, anxiety symptoms, hostility, phobic-anxiety, and paranoid tendency. Additional symptoms include vegetative and other clinical indicators. The BSRS is composed of 30 items rated on the basis of degree of distress caused by that item over the past week. Each dimension is assessed by several questions with a 5-point Likert scale (0-4 points). The severity of a psychopathologic factor is expressed with an index calculated from the sum of scores divided by the number of questions in that specific dimension. The General Symptom Index (GSI), a mean score of all BSRS items, represents the global severity of psychological distress (PD), and a higher GSI indicates more severe PD. The BSRS has been reported to be a reliable and valid psychiatric self-rating scale for use in psychosomatic research.

SECONDARY OUTCOMES:
Bladder wall blood flow | 12 hours
  vascularization index (VI) 、flow index (FI) and vascularization flow index (VFI)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan